CLINICAL TRIAL: NCT00976430
Title: To Study the Safety and Efficacy of Bone Marrow Derived Mesenchymal Stem Cells Transplant in Parkinson's Disease
Brief Title: Autologous Mesenchymal Stem Cell Transplant for Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Adequate no. of patients could not be recruited in the set time frame.
Sponsor: Jaslok Hospital and Research Centre (Other)
Responsible Party: Principal Investigator, Dr Paresh Doshi, In-charge Stereotactic and Functional neurosurgery, Jaslok Hospital and Research Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JHC525
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
Keywords: Autologous Stem Cells.
MeSH Terms: conditions — Parkinson Disease | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapy for Parkinson's disease (Experimental): Stem cell derived from the bone marrow of the patient will be stereotactically transplanted in the striatum.These stem cell are the expected to grow up into dopamine secreting neural cells.
  Interventions: Procedure: Autologous Bone marrow derived stem cells transplant

INTERVENTIONS:
Procedure: Autologous Bone marrow derived stem cells transplant — Stem cells are derived from the bone marrow of the patient and processed at Reliance life sciences.The stem cells are the stereotactically implanted in the striatum.
  Other Names: stem cells; cell therapy for Parkinson's disease

SUMMARY:
This study is intended to look at the safety and efficacy of the use of autologous bone marrow derived stem cell transplant in patients with advanced Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease, a neurodegenerative disorder, still at its best can only be controlled by medical or surgical treatment. For more than two decades various groups have tried using modified cell transplants for curing this disease. Earlier results with use of fetal mesencephalic cell transplant were encouraging, but this had to be discontinued due to severe side effects.

Current interest, in the use of Mesenchymal stem cells as a pluripotent cell for developing neural cells has been the background for this study. Reliance Life sciences had found encouraging results with the use of human MSCs in Rat model of PD. Based on this and other data, Jaslok Hospital and Research Centre has initiated a pilot study to investigate the efficacy of Autologous MSCs in treating advanced PD. This cells will be harvested from bone marrow, processed at RLS laboratory and transplanted by stereotactic techniques into the striatum of the patient.

ELIGIBILITY:
Inclusion Criteria

* Male or female between 35-70 years of age.
* Patient with current diagnosis of PD with motor complications (as confirmed by neurologist) as per the standard criteria and guidelines.
* Patients with at least 5 years since the disease.
* Responsiveness to Levodopa or dopa agonist. This is defined as improvement between Off and On UPDRS by at least 33% of the Motor UPDRS.
* PD of Stage 2.5, 3 & 4 of HOEHN & YAHR staging.
* Stable Parkinsonian medications for the 60 days prior to the surgical therapy.
* MRI not showing gross atrophy or any other pathology of brain.
* Patients with score less than 19 for the Montgomery-Asberg Rating Scale (MADRS) for Depression.
* NO Significant cognitive impairment.MMSE > 24.
* The participant is able to comply with and understand the required visit schedule and all required tests and procedures.
* The participant (and/or LAR) must sign an informed consent.

Exclusion Criteria:

* History of intracranial surgeries or implantation of a device for Parkinson's disease two years prior to treatment.
* History of psychiatric disorders like schizophrenia or psychotic disorders.
* History of other malignancy, with the exception of treated cutaneous squamous cell or basal cell carcinoma, within 5 years.
* Contraindication for MRI
* General medical contraindications for surgery like coagulopathy
* Subjects with abnormal hematology and chemistry values, unless the out of range values are clinically significant with respect to general surgery.
* Severe skin infection or osteomyelitis at the site of bone marrow aspiration potentially limiting the procedure.
* Positive test results for HIV.
* History of drug or alcohol abuse
* Pregnant or nursing women

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement in clinical condition of the patient assessed using UPDRS (UNIFIED PARKINSON'S DISEASE RATING SCALE) and Time Tests. | Up to 18 months from the day of stem cell transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Paresh k Doshi, MCh, Principal Investigator — Incharge Stereotactic and functional Neurosurgery,Jaslok Hospital and Research Centre.
Locations (1):
- Jaslok Hospital And Research Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arias-Carrion O, Yuan TF. Autologous neural stem cell transplantation: a new treatment option for Parkinson's disease? Med Hypotheses. 2009 Nov;73(5):757-9. doi: 10.1016/j.mehy.2009.04.029. Epub 2009 May 24. PMID 19467573